CLINICAL TRIAL: NCT04546607
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel, Study Assessing NuvastaticTM (C5OSEW5050ESA) 1000 mg (3 Times a Day) in Improving Fatigue in Patients With Solid Stage I - IV Tumors
Brief Title: Evaluation of Clinical Efficacy and Safety of Nuvastatic in Cancer Asthenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Natureceuticals Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBSB0045011CRA
Record Dates: First submitted 2020-05-11; First posted 2020-09-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Asthenia; Cancer
MeSH Terms: conditions — Asthenia; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial. the study was intervention type, in which different cancer patients were administered with relevant chemotherapeutic drugs + Nuvastatic. The drug-type of Nuvastatic is a botanical drug which was used as chemo-adjuvant.
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuvastatic TM (Experimental): Nuvastatic TM (C5OSEW5050ESA) capsule 1000 mg administered orally 3 times a day for 9 weeks.
  Interventions: Other: Nuvastatic TM (C5OSEW5050ESA) 1000 mg
- Placebo (Placebo Comparator): Excipient, without Nuvastatic TM (C5OSEW5050ESA) capsule administered orally 3 times a day for 9 weeks.
  Interventions: Other: Nuvastatic TM (C5OSEW5050ESA) 1000 mg

INTERVENTIONS:
Other: Nuvastatic TM (C5OSEW5050ESA) 1000 mg — Nuvastatic TM is a patented polymolecular botanical medicine made from Lanctos 75TM which is a proprietary high potency herbal standardized extract.

SUMMARY:
Nuvastatic TM (C5OSEW5050ESA)is a special formulation derived from the standardized extract of O. stamineus leaves developed by Natureceuticals Sdn. Bhd. The extract is prepared from meticulous extraction using sophisticated phytochemical techniques, where the particular phytopharmaceuticals (active ingredients) are being concentrated to achieve the desired therapeutic efficacy. In the proposed human study, it is anticipated that administering dietary supplement of standardized O. stamineus rosmarinic acid-enriched Nuvastatic TM (C5OSEW5050ESA) 1000 mg (3 times a day), can ameliorate fatigue in cancer patients. This is based on scientific studies that support its ability in reducing oxidative damage and restore mitochondrial and other cellular functions involved in cellular energy production. It is further hypothesized that the anti-inflammatory, antinociceptive anti-oxidant, and neuroprotective properties of the active compound rosmarinic acid may also potentially assist in pain control, sleep loss, lethargy and other symptoms strongly associated with cancer-related fatigue.

DETAILED DESCRIPTION:
All stage I-IV solid tumors patients are planned to receive or already receiving chemotherapy or radiotherapy including palliative chemotherapy and radiotherapy meeting the eligibility criteria will be consented and pre-screened for fatigue using Brief Fatigue Inventory (BFI). Subjects will be administered a BFI questionnaire prior to the commencement of their chemotherapy (preferably 1st chemotherapy cycle) or radiotherapy treatment.

Patients will be assessed again using the BFI questionnaire on day 1 of their next chemotherapy cycle or the following week of radiotherapy. Patients will not be considered for study enrolment if the fatigue severity does not increase by at least one score from the previous assessment during the pre-screening. Those with newly developed fatigue or worsening of their fatigue score (i.e. from moderate to severe, mild to moderate, or mild to severe) will be consented for study enrolment. The subject who signed informed consent, pre-screened and is subsequently eligible for study enrolment/randomization will be enrolled into either Nuvastatic TM or Placebo group

ELIGIBILITY:
Inclusion Criteria:

Males or females, ≥ age 18 Patients with solid tumors, Stage I-IV Patients who received, receiving, or plan to receive chemotherapy and/or ≥ 1 week of radiotherapy.

ECOG 0-2 Life expectancy ≥ 6 months Ability and willingness to provide written informed consent and comply with study requirement

Exclusion Criteria:

1. Known allergy to Nuvastatic TM (C5OSEW5050ESA) or any of the excipient used in the preparation of the investigational product 2. Any other known existing condition that contraindicates with the use of investigational product 3. Inability to take or consume the investigational product per protocol-specified route of administration including peptic ulcer disease, chronic gastritis, hypotension, and systolic blood pressure <90mmgHg.
2. Inability to understand local language (s) for which BFI, EORTC-QLQ- C30, FACIT-F, visual analogue scale for fatigue questionnaire 5. Any condition (e.g. Psychological, geographical, etc.) that does not permit compliance with the study or follow up procedures 6. Participation in any other clinical study using an investigational medicinal product or device within 28 days prior to baseline visit 7. Treatment with medications or supplements frequently associated with fatigue, such as interferon (within the last four months), beta-blockers, calcium channel blockers, benzodiazepines, sedating antihistamines, antidepressants, antipsychotics, or melatonin. In select instances, patients using these medications may be enrolled if, in the opinion of the investigators, their fatigue is clearly unrelated to the medication.
3. Untreated or uncontrolled comorbidities that influence fatigue, including thyroid disorders (TSH> 5 mcIU/mL), anemia (Hemoglobin< 9 g/dL), major depression, active substance abuse, or other conditions as determined by the enrolling physician. Comorbidities that are adequately controlled will not exclude patients.
4. Chronic renal failure patients with raised serum potassium levels and abnormal renal function 10. Untreated sleep disorders such as obstructive sleep apnea or restless leg syndrome 11. Decompensated cirrhosis (encephalopathy, gastrointestinal bleeding, ascites, bilirubin > 2) within the last six months 12. Patients planning to travel outside the time zone during the study period 13. Known or suspected significant gastrointestinal motility disorder, obstruction, or structuring disease 14. Severe malnutrition according to WHO criteria. 15. Upon examination, the patients may be deemed to have any of the following conditions:

   a. Bipedal edema b. Visible severe wasting c. Weight for height more than 3 standard deviations below the median of international reference population d. Fever related to systemic infection (especially Gram-negative coliforms such as Escherichia coli and Klebsiellapneumoniae), neutropenic sepsis e. Respiratory distress f. Heart failure g. Electrolyte abnormalities (hypophosphataemia, hypokalemia/ hyperkaliemia, hypoglycemia, etc.) h. Marked anorexia i. Profuse diarrhea j. Shock
5. The patient is female and is pregnant or fertile and is not practicing adequate methods of contraception, is planning to become pregnant within 1 month of the study, is breastfeeding. Note: Females who are breastfeeding should not be discouraged from breastfeeding for the sole purpose of enrolling in the study. Females who choose to defer breastfeeding until 5 days after the last dose of study drug to allow the elimination of the drug from breast milk will be eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Improving Fatigue in Patients with Solid Stage I - IV Tumors. | Measured at baseline (Visit 2) (week 2)
  Functional Assessment of Chronic Illness Therapy Fatigue FACIT-F scale as primary endpoint. FACIT-Fatigue Scale: (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much)
To evaluate efficacy of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Improving Fatigue in Patients with Solid Stage I - IV Tumors. | Measured at Visit 3 (week 3)
  Functional Assessment of Chronic Illness Therapy Fatigue FACIT-F scale as primary endpoint. FACIT-Fatigue Scale: (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much)
To evaluate efficacy of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Improving Fatigue in Patients with Solid Stage I - IV Tumors. | Measured at Visit 6 (week 6)
  Functional Assessment of Chronic Illness Therapy Fatigue FACIT-F scale as primary endpoint. FACIT-Fatigue Scale: (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much)
To evaluate efficacy of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Improving Fatigue in Patients with Solid Stage I - IV Tumors. | Measured at Visit 9 (week 9)
  Functional Assessment of Chronic Illness Therapy Fatigue FACIT-F scale as primary endpoint. FACIT-Fatigue Scale: (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much)
To evaluate the safety and tolerability of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Patients with Solid Stage I - IV Tumors. | Measured at baseline (Visit 2) (week 2)
  Visual Analogue fatigue scale (VAFS) as primary endpoint. Fatigue with 0 being worst and 10 being normal.
To evaluate the safety and tolerability of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Patients with Solid Stage I - IV Tumors. | Measured at Visit 3 (week 3)
  Visual Analogue fatigue scale (VAFS) as primary endpoint. Fatigue with 0 being worst and 10 being normal.
To evaluate the safety and tolerability of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Patients with Solid Stage I - IV Tumors. | Measured at Visit 6 (week 6)
  Visual Analogue fatigue scale (VAFS) as primary endpoint. Fatigue with 0 being worst and 10 being normal.
To evaluate the safety and tolerability of CANSSUFIVE® Nuvastatic (C5OSEW5050ESA) in Patients with Solid Stage I - IV Tumors. | Measured at Visit 9 (week 9)
  Visual Analogue fatigue scale (VAFS) as primary endpoint. Fatigue with 0 being worst and 10 being normal.

SECONDARY OUTCOMES:
Quality of Life (QoL) | Measured at baseline (visit 2) (week 2), visit 3 (week 3), visit 4 (week 6), and visit 5 (week 9).
  Overall QoL improvement using EORTC-QLQ-C30. Scale 1 (worse) to 10 (better).
Fatigue Severity Scale | Measured at baseline (visit 2) (week 2), visit 3 (week 3), visit 4 (week 6), and visit 5 (week 9).
  Fatigue Severity Scale (FSS). Scale ranging from 1 ("strongly disagree") to 7 ("strongly agree").
Brief Fatigue Inventory | Measured at baseline (visit 2) (week 2), visit 3 (week 3), visit 4 (week 6), and visit 5 (week 9).
  Brief Fatigue Inventory. 11-point rating scale developed to assess subjective fatigue. Fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels.
Vitality subscale of the Medical Outcome Scale Short Form-36 (SF-36) | Measured at baseline (visit 2) (week 2), visit 3 (week 3), visit 4 (week 6), and visit 5 (week 9).
  Vitality subscale of the Medical Outcome Scale Short Form-36 (SF-36). Scale ranging from 0 (worst possible health state) to 100 (best possible health state).
F2-isoprostane | Measured at baseline (visit 2) (week 2), visit 3 (week 3), visit 4 (week 6), and visit 5 (week 9).
  urinary F2-isoprostane as a biomarker for fatigue reduction
The adverse events | During 9 weeks intervention and at end of intervation on 9th week.
  The occurrence and severity of adverse effects are measured by a severity score scale and system organ class (gastrointestinal disorders, general disorders, and administration site conditions, nervous system disorders) in treatment vs placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Ghanashyam Biswas, PHD, Principal Investigator — Sparsh Hospitals & Critical Care Pvt. Ltd.
Locations (1):
- Notrox Research Pvt Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng ML, Majid AMSA, Yee SM, Natesan V, Basheer MKA, Gnanasekaran A, Al-Suede FSR, Parish C, Dalal M, Ming LC, Nazari V M, Khan SS, Stn Hameed Sultan SB, Babu KG, Majid ASA, Abdul Aziz MAS. A phase II randomized, double-blind, placebo-controlled study of Nuvastatic (C50SEW505OESA), a standardized rosmarinic acid-rich polymolecular botanical extract formulation to reduce cancer-related fatigue in patients with solid tumors. Support Care Cancer. 2024 May 6;32(6):331. doi: 10.1007/s00520-024-08536-w. PMID 38710920